CLINICAL TRIAL: NCT03878888
Title: The Use of Exparel (Liposomal Bupivacaine) for Bilateral TAP (Transversus Abdominis Plane) Blocks in Open Abdomen Surgery for Postoperative Pain Control
Brief Title: Exparel Use in Bilateral TAP Blocks for Postoperative Pain Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Luke's Hospital, Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: stluke
Record Dates: First submitted 2019-03-09; First posted 2019-03-18 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Postoperative Pain; Surgery; Anesthesia, Local
Keywords: liposomal bupivacaine; TAP block; pain control
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Injections

STUDY DESIGN:
Intervention Model Description: experimental group: patients having open abdominal surgery that will receive a bilateral TAP block with Exparel control group: patients having open abdominal surgery that will not receive a bilateral TAP block with Exparel
Masking Description: no masking; will provide qualified patients the opportunity to receive Exparel (liposomal bupivacaine) in Bilateral TAP blocks for open abdomen surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Exparel use in TAP block (Experimental): Exparel used in bilateral TAP block for open abdomen surgery
  Interventions: Drug: Exparel 266 MG Per 20 ML Injection
- no TAP block (No Intervention): these patients, N=20, did not received a bilateral TAP block for postoperative pain control. Instead, pain control involves PO/IV pain medications

INTERVENTIONS:
Drug: Exparel 266 MG Per 20 ML Injection — patients receive Exparel in bilateral TAP blocks for open abdomen surgery
  Other Names: liposomal bupivacaine
  Arms: Exparel use in TAP block

SUMMARY:
To determine if Exparel (Liposomal Bupivacaine, an FDA approved drug) use in ultrasound guided Transversus Abdominis Plane (TAP) blocks may reduce opioid requirement use postoperatively, reduce pain scores postoperatively, reduce incidence of nausea in the postop period, and decrease length of hospital stay

DETAILED DESCRIPTION:
Exparel is liposomal form of bupivacaine, a local anesthetic. Secondary to its liposomal nature, Exparel slowly releases bupivacaine into the area injected (ultrasound guided field block) so that it may provide relief from pain for up to 48-72 hours time.

Exparel in TAP blocks may be performed on patients undergoing open or laparoscopic hand assisted abdomen/pelvic procedures, who are NOT candidates for an epidural (anticoagulation medication use, history of spine surgery with metal hardware of the mid-lower back) or as a rescue block for patients who undergo laparoscopic surgery but converted to open abdominal surgery in the operating room.

This block is usually performed intraoperatively (before patient wakes up from anesthesia) or in the immediate postop recovery unit (PACU) area.

Anesthesia personnel who have been well trained to perform ultrasound guided bilateral TAP blocks will combine Exparel 20 cc's with 0.25% Bupivicaine 20 ccs and 20 ccs of normal saline into a 60 cc syringe. With ultrasound machine, they will locate the TAP block on each side of abdomen with a Stimuplex needle. Once the TAP area is found, hydrodissection with normal saline is used to confirm TAP area, and then 30 ccs of the Exparel/0.25% Bupivacaine/normal saline solution administered to each side.

Patients are seen in the PACU area, where pain scores and oral morphine equivalents (OME) are calculated. Patient seen in postoperative day (POD) 1 to discuss expectations of pain control and goals for pain management (i.e. use of multimodal pain regimen and goals to decrease opioid use). A flyer (approved by the Patient Education Committee) is provided to patient on POD 1 for further patient education. Pain scores and OMEs calculated for POD 0-5. Progress notes in patient's chart and patient interview also discloses if patient had episodes of N/V, another data point we will collect. We will finally review patient charts for length of admission (date of admission to date of discharge) Our control group: patients that had open abdominal or hand assisted laparoscopic surgery and who did not receive a TAP block, and received mainly opioids for postop pain control. For the comparison (control) group, we will calculate OME requirements while in PACU, and from POD 1-POD 5. We will see patients during POD 1 to discuss expectations of pain control and goals for pain management. Progress notes in patient's chart and patient interview also discloses if patient had episodes of N/V, another data point we will collect. We will finally review patient's chart for length of admission (date of admission to date of discharge) We are looking for an N=20 for the Exparel TAP block (experimental) group and N=20 for no TAP block (control) group

ELIGIBILITY:
Inclusion Criteria:

* Women of Reproductive Potential
* Men of Reproductive Potential
* Minorities
* Healthy Controls/Volunteers
* Employees/Students
* Vulnerable populations (trauma victims, students > 18 yrs age, aged infirm, substance abusers, impoverished, terminally ill,)

patients of above inclusion criteria who 1) are not candidates of an neuraxial blockade (i.e. epidural) for postoperative pain control 2) who underwent a laparoscopic to open procedure intraoperatively

Exclusion Criteria:

* advanced dementia, not oriented to time or place
* advanced liver disease
* pregnant patients
* allergy to amide local anesthesia
* allergy to methemoglobinemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Reduce opioid requirement use (calculated oral morphine equivalents (OME)) for 2-3 days time after surgery. | up until postoperative day 5
  will review opioid/narcotic use in patient's chart
Reduce pain scores after surgery | up until postoperative day 5
  Numerical Rating Scale: 0-10; 0 being no pain, 10 being worst pain imaginable possible

SECONDARY OUTCOMES:
Reduce incidence of nausea postoperatively | up until Postoperative day 5
  will review in daily progress notes incidence of nausea
Decrease length of hospital stay | up until postoperative day 5
  will review patient's admission encounter in chart and see when patient is discharged

CONTACTS AND LOCATIONS:
Overall Officials: Anna Ng Pellegrino, MD, Principal Investigator — St. Luke's University Health Network - Anesthesia
Locations (1):
- St. Luke's University Hospital Health Network, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seagle BL, Miller ES, Strohl AE, Hoekstra A, Shahabi S. Transversus abdominis plane block with liposomal bupivacaine compared to oral opioids alone for acute postoperative pain after laparoscopic hysterectomy for early endometrial cancer: a cost-effectiveness analysis. Gynecol Oncol Res Pract. 2017 Aug 22;4:12. doi: 10.1186/s40661-017-0048-7. eCollection 2017. PMID 28852531
- [Result] Fayezizadeh M, Majumder A, Neupane R, Elliott HL, Novitsky YW. Efficacy of transversus abdominis plane block with liposomal bupivacaine during open abdominal wall reconstruction. Am J Surg. 2016 Sep;212(3):399-405. doi: 10.1016/j.amjsurg.2015.12.026. Epub 2016 Apr 12. PMID 27156796
- [Result] Feierman DE, Kronenfeld M, Gupta PM, Younger N, Logvinskiy E. Liposomal bupivacaine infiltration into the transversus abdominis plane for postsurgical analgesia in open abdominal umbilical hernia repair: results from a cohort of 13 patients. J Pain Res. 2014 Aug 16;7:477-82. doi: 10.2147/JPR.S65151. eCollection 2014. PMID 25170277
- [Result] Gorfine SR, Onel E, Patou G, Krivokapic ZV. Bupivacaine extended-release liposome injection for prolonged postsurgical analgesia in patients undergoing hemorrhoidectomy: a multicenter, randomized, double-blind, placebo-controlled trial. Dis Colon Rectum. 2011 Dec;54(12):1552-9. doi: 10.1097/DCR.0b013e318232d4c1. PMID 22067185
- See also: Ching, Heidi. A comparison of Exparel to Bupivacaine in TAP block for Abdominal Gynecologic surgery. clinicaltrials.gov : NCT03304444. — http://clinicaltrials.gov
- See also: Turan Et. Al. Bilateral Transversus Abdominis Plane Block with Exparel vs. Continuous Epidural Analgesia with Bupivacaine. Clinical trials.gov: NCT02996227 — http://clinicaltrials.gov